CLINICAL TRIAL: NCT04690686
Title: Open-Label Study Evaluating the Safety and Effectiveness of Immunopheresis With the LW-02 Column Alone or in Combination With Paclitaxel or Atezolizumab in Removing Soluble Tumor Necrosis Factor Receptors to Treat Patients With Advanced, Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Immunopheresis Alone or in Combination With Paclitaxel or Atezolizumab in Non-small Cell Lung Cancer (NSCLC).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunicom Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP7-008
Record Dates: First submitted 2020-10-23; First posted 2020-12-31 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Open-label, phase 2a pilot study of Immunicom's LW-02 column-combined with low-dose chemotherapy or immunotherapy.
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LW-02 device immunopheresis combined with atezolizumab (Experimental): LW-02 column immunopheresis treatments ~3x/week for 16 weeks plus atezolizumab 1200 milligrams (mg) q3w until disease progression or loss of clinical benefit, death, unacceptable toxicity, withdrawal of consent, or study termination by sponsor, whichever occurs first [N=8]
  Interventions: Device: LW-02 device immunopheresis combined with atezolizumab
- LW-02 device immunopheresis combined with weekly paclitaxel (Experimental): LW-02 column immunopheresis treatments ~3x/week for 16 weeks plus paclitaxel 80 mg/m2 /week × 6 followed by 2 weeks rest until disease progression, death, unacceptable toxicity, withdrawal of consent, or study termination by sponsor, whichever occurs first. [N=8]
  Interventions: Device: LW-02 device immunopheresis combined with weekly paclitaxel
- LW-02 device immunopheresis (Experimental): LW-02 column immunopheresis treatments ~3x/week for 16 weeks alone until disease progression, death, unacceptable toxicity, withdrawal of consent, or study termination by sponsor, whichever occurs first. [N=8]
  Interventions: Device: LW-02 device immunopheresis

INTERVENTIONS:
Device: LW-02 device immunopheresis combined with atezolizumab — The LW-02 device comprises an immunoadsorption affinity column, employing a proprietary human recombinant protein, single chain TNF-α ligand, covalently linked to a bead resin, that both enhances the capture efficiency of sTNF-Rs while avoiding complications from column leaching. Reduced sTNF-R plasma levels may lead to objective tumor responses. In combined treatment arm the immunopheresis procedure is combined with standard dose immunotherapy (atezolizumab) to potentially enhancing its cytotoxic effect.
  Other Names: Plasma soluble TNF receptor pulldown + immunotherapy.
  Arms: LW-02 device immunopheresis combined with atezolizumab
Device: LW-02 device immunopheresis combined with weekly paclitaxel — The LW-02 device comprises an immunoadsorption affinity column, employing a proprietary human recombinant protein, single chain TNF-α ligand, covalently linked to a bead resin, that both enhances the capture efficiency of sTNF-Rs while avoiding complications from column leaching. Reduced sTNF-R plasma levels may lead to objective tumor responses. In combined treatment arm the immunopheresis procedure is combined with low dose chemotherapy to potentially enhancing its cytotoxic effect.
  Other Names: Plasma soluble TNF receptor pulldown + chemotherapy
  Arms: LW-02 device immunopheresis combined with weekly paclitaxel
Device: LW-02 device immunopheresis — The LW-02 device comprises an immunoadsorption affinity column, employing a proprietary human recombinant protein, single chain TNF-α ligand, covalently linked to a bead resin, that both enhances the capture efficiency of sTNF-Rs while avoiding complications from column leaching. Reduced sTNF-R plasma levels may lead to objective tumor responses.
  Other Names: Plasma soluble TNF receptor pulldown
  Arms: LW-02 device immunopheresis

SUMMARY:
This pilot study aims to evaluate the short-term and long-term safety, tolerability, and effectiveness of immunopheresis with the LW-02 column in removal of sTNFRs from plasma of patients with advanced, refractory NSCLC and to detect a potential disease control signal when employed in combination with low dose chemotherapy (ie, paclitaxel), immunotherapy (ie, atezolizumab) in patients who already failed first-line therapy, or as monotherapy in patients who already have failed second-line therapy.

DETAILED DESCRIPTION:
This is an open-label, Phase 2a pilot study of Immunicom's LW-02 column- combined with low-dose chemotherapy or immunotherapy in patients who have failed first-line treatment or employed as monotherapy in patients who have failed second-line therapy-to evaluate the short-term and long-term safety, tolerability and effectiveness of these approaches in removing sTNF-Rs and the potential for disease control in advanced, refractory NSCLC patients. Along with LW-02 column immunopheresis, patients enrolled in Arm 1 will receive combination immunotherapy with atezolizumab and patients enrolled in Arm 2 also will receive combination chemotherapy with paclitaxel. Patients in Arm 3 will be treated with LW-02 column immunopheresis alone as a third-line treatment regimen, assuming the first-line treatment included a platinum salt. Following study qualification, patients will be assigned to the appropriate treatment. All patients may receive up to 48 LW-02 column-based immunopheresis treatments over a 16-week (4-month) period with up to 3 treatments per week). Importantly, each LW-02 immunopheresis treatment should last up to 3 hours and process, approximately, 2 times the patient's plasma volume (2PV).

Each patient assigned to the treatment with LW-02 column-based immunopheresis will require central vascular access for the procedure. In general, a cuffed, tunneled dual-lumen catheter will be inserted into a central vein and remain in situ throughout the 16-week treatment phase (or longer if additional treatment is clinically indicated). The catheter will be used to connect the inlet and return lines of the apheresis system to the patient. Immunopheresis treatments will be performed using the LW-02 column used inline with a centrifugal apheresis system that allows for secondary plasma processing system (eg, the Terumo BCT Spectra Optia Apheresis System® or alternate apheresis system). Proper anticoagulation of the centrifugal apheresis device is generally provided by utilizing acid citrate dextrose formula A (ACD-A).

Patients will be followed and clinically evaluated for two-years posttreatment. In Year 1, patients will be clinically evaluated at 3, 6, 9, and 12 months from the end-of-treatment (EOT) visit. In Year 2 quarterly (every 3 months) telephone contacts will be made to determine overall survival.

ELIGIBILITY:
This pilot study will enroll 24 patients with measurable advanced, refractory NSCLC (incurable stage IIIB and stage IV) histologically confirmed as squamous or adenocarcinoma following failure of:

* 1st standard line of systemic treatment that included a platinum salt administered in a palliative setting (Arms 1 and 2); or,
* 2nd line standard chemotherapy assuming the first line included a platinum salt (Arm 3). Inclusion criteria are to be confirmed within 28 days of the first LW-02 immunopheresis treatment (preferably as proximate to the date of the first treatment as possible):

  1. Signed Informed Consent Form
  2. Age 18 - 75 years of age
  3. Able to comply with the study protocol in the investigator's judgment
  4. Histologically or cytologically documented stage IIIb or stage IV squamous or adenocarcinoma NSCLC that has progressed despite 1 line of chemotherapy that included a platinum salt (Arms 1 and 2) or 2 lines of standard chemotherapy assuming the 1st line included a platinum salt (Arm 3). [Patients with adenocarcinoma must have confirmed negative status of EGFR gene mutation and ALK fusion gene and ROS1.]
* Patients who discontinued previous treatments (first- or second-line) due to intolerance are also eligible.
* Staging must be according to the UICC/AJCC system, 7th edition (Detterbeck et al. 2009)
* Pathological characterization may be conducted on tumor specimens from earlier stage disease, but the tumor samples must have been sufficient to confirm squamous or adenocarcinoma histologically
* Combined radiation/chemotherapy treatment (chemoradiation) counts as one prior chemotherapy regimen if < 6 months have elapsed between the last dose and the date of recurrence
* Adjuvant/neoadjuvant chemotherapy is not counted as a line of treatment except for cases where the relapse is diagnosed < 6 months from the end of adjuvant/neoadjuvant chemotherapy that included a platinum salt.
* Debulking surgery and anticancer agents used for pleurodesis are not counted as lines of therapy 5. Must be able to provide archival pathological material from primary or metastatic site (formalin-fixed paraffin embedded [FPPE] tissue block) for central NSCLC confirmation and verification of NSCLC subtype and tmTNF expression 6. Body mass ≥ 35 kg 7. Life expectancy of at least 3 months with malignancy; expected to live for one year without malignancy. 8. Adequate organ function:

  1. Hemoglobin ≥ 9.5g/dL (may be achieved with transfusion support)
  2. Absolute Neutrophil Count (ANC) ≥1.5 × 109/L (without granulocyte colony-stimulating factor support within 2 weeks prior to the first study treatment)
  3. Platelets (PTL) ≥ 100 × 109/L
  4. AST/ALT ≤2.5×ULN (patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN; patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 × ULN)
  5. Serum creatinine (S-Cr) ≤ 1.2 ULN
  6. Albumin ≥ LLN
  7. Bilirubin ≤ 1.5 ULN
  8. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. This applies only to patients who are not receiving therapeutic anticoagulation agents.
  9. Patients should not be receiving therapeutic anticoagulation. Prophylactic low doses of ASA are acceptable.
  10. Serum calcium level within normal range. 9. The last dose of prior systemic anticancer therapy must have been administered

      * 14 days prior to study treatment initiation assuming all substantial chemotherapy toxicities recovered satisfactorily. 10. Having not used antibiotics in the last month prior the start of the screening or, at least, prior to obtaining a baseline microbiome sample. 11. Measurable disease, as defined by RECIST v1.1 12. Patients with asymptomatic CNS metastases (treated or untreated), as determined by CT or MRI evaluation during screening and prior radiographic evaluation, are eligible if do not require corticosteroids dose adjustments due to in the last 4 weeks.

        13. ECOG performance status 0, 1 or 2. 14. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use double barrier contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 5 months after the last treatment.

        15. Patients must have recovered (i.e., improvement to Grade 1 or better) from all acute toxicities from previous therapy, excluding alopecia.

Exclusion criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Symptomatic CNS metastases
2. Leptomeningeal disease
3. Uncontrolled pericardial effusion or ascites requiring recurrent drainage procedures
4. Previous use of paclitaxel (not applicable for patients enrolled in Arm 3).
5. Pregnant or lactating or intending to become pregnant during the study or for at least 5 months after the least study treatment. Women who are not postmenopausal (postmenopausal defined as ≥ 12 months of non-drug-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 2 weeks prior to initiation of study treatment
6. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome)
7. Significant cardiovascular disease, such as New York Heart Association cardiac disease ≥ Class III, myocardial infarction within 3 months, unstable arrhythmias, or unstable angina
8. Patients with known coronary artery disease or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
9. Patient with known persistent, uncontrolled hypotension
10. Significant renal disorder requiring dialysis or indication for renal transplant
11. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to study treatment initiation
12. Major surgical procedure within 4 weeks prior to study treatment initiation or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
13. Fever, or any active immunosuppressive systemic infection including history of human immunodeficiency virus (HIV) infection
14. Other serious diseases (e.g., life expectancy less than 3 months) including active second malignancy except for basal cell carcinoma or cervical carcinoma in situ
15. Active infection
16. Patients in whom vascular access is not considered achievable
17. Use of any standard high dose or low dose chemotherapy or immunosuppressive therapies and or standard radiation therapy concurrently as well anticipated need for any of the former during the study
18. Body mass index (BMI) ≥ 35 kg/m2
19. Any condition that the patient's physician determines to be detrimental to the patient participating in this study; including any clinically important abnormal clinical laboratory values or concurrent medical events
20. Inability to understand the local language affecting the use of the patient QOL instruments.
21. Need for regular treatment with an angiotensin converting enzyme (ACE) inhibitor during the study; patients should discontinue treatment at least 14 days prior to the first LW-02 column immunopheresis treatment.

Additional exclusions for patients to be treated in Arm 1 (with atezolizumab):

1. Previous use of atezolizumab.
2. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
3. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
4. History of autoimmune disease is allowed if controlled and on stable treatment (i.e., same treatment, same dose) for the last 12 weeks, with the exception of:

   1. Patients taking concurrent abatacept or belatacept treatment (prior therapy must have been withdrawn for > 8 weeks)
   2. Patients with a history of serious or life threatening immune-related events
   3. No more than 1 concomitant autoimmune disease at the time of study entry is allowed unless one of them is:

   i. Autoimmune-mediated hypothyroidism on a stable dose of thyroid replacement hormone ii. Controlled Type I diabetes mellitus on a stable dose of insulin regimen iii. A medical history of such entities as atopic disease or childhood arthralgia, where the clinical suspicion of autoimmune disease is low. In addition, transient autoimmune manifestations of an acute infectious disease that resolved upon treatment of the infectious agent are not excluded (eg, acute Lyme arthritis) iv. Vitiligo.
5. Prior allogeneic stem cell or solid organ transplantation
6. History of idiopathic pulmonary fibrosis, including pneumonitis, drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan

   a. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
7. Active tuberculosis

   a. In patients who have a potentially high likelihood of latent tuberculosis (e.g., recent contact with an infectious carrier, residence in a locale with high TB burden), absence of Mycobacterium tuberculosis infection must be confirmed before enrollment according to local practice standards
8. Administration of a live, attenuated vaccine within 4 weeks prior to study treatment initiation

   1. Influenza vaccination should be given during influenza season only (e.g., approximately October to March in the Northern Hemisphere).
   2. Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to study treatment initiation or at any time during the study.
9. Prior treatment with CD137 agonists or immune checkpoint blockade therapies other than anti-PD-1 therapy, including anti-PD-L1 therapeutic antibodies
10. Treatment with systemic immunostimulatory agents (including, but not limited to, interferons or interleukin 2) within 4 weeks or five half-lives of the drug, whichever is longer, prior to initiation of study treatment

    a. Prior cancer vaccines and cellular immunotherapy are permitted
11. Specifically for patients without autoimmune disease: treatment with systemic corticosteroids or other systemic immunosuppressive medications including, but not limited to: prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents within 2 weeks prior to study treatment initiation, or anticipated requirement for systemic immunosuppressive medications during the trial

    1. For patients with CNS metastases and lung cancer related dyspnea, use of prednisone at a stable dose (or dose equivalent) of ≤ 20 mg/day is acceptable.
    2. The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (eg, fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency and topical steroids for cutaneous diseases are allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 16 weeks
  Treatment-Emergent Adverse Events which will be analysed in study ill be:
  1. Adverse Event (AE)
  2. Serious Adverse Events (SAE)
  3. Adverse Device Effect (ADE)
  4. Serious Adverse Device Effect (SADE) Each of the Treatment-Emergent Adverse Events will be assessed for their seriousness, severity [using NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 v. 5.0] and causality (relationship with the use of the investigated medical device).
Column performance effectiveness | 16 weeks
  Column efficiency and effectiveness in removal of sTNF-Rs from patient plasma without clinically-meaningful leaching of capture ligand (SC-TNF-α) - change in sTNF-R and TNF-α plasma levels from initiation to the end of each
  LW-02 column perfornance effectiveness will be assessed to measure over 30 minutes (sTNF-Rs) and over the duration (leaching) of each procedure, respectively:
  * Removal of soluble TNF receptor 1 (sTNF-R1)
  * Removal of soluble TNF receptor 2 (sTNF-R2)
  * Leaching of sc-TNF-α from the column
Incidence of Treatment-Emergent Adverse Events of special interest. | 16 weeks
  Incidence of Treatment-Emergent Adverse Events of special interest assessment will include:
  1. tumor lysis syndrome and
  2. systemic inflammatory response syndrome. These events may or may not be serious and they may or may not be considered related to study treatment. Regardless of relationship or severity, these events will be recorded if they start after the first application of study treatment and will be followed until resolution.

SECONDARY OUTCOMES:
Patient functioninig with Eastern Cooperative Oncology Group (ECOG) | 16 weeks
  Eastern Cooperative Oncology Group (ECOG) scale describes patient's functioning in terms of ability to care for themselves, daily activity, and physical ability (walking, working). The scale grades 0 to 5 (0=fully active while and 5=dead).
Quality of life assessment with EQ-5D-5L scale | 16 weeks
  EQ-5D-5L scale to assess: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels:
  from no problems to extreme problems.
Quality of life assessment with EORTC-QLQ-C30 scale | 16 weeks
  EORTC-QLQ-C30 scale measures cancer patients' physical, psychological and social functions. The EORTC QLQ-C30 comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Quality of life assessment with EORTC-QLQ-LC29 scale | 16 weeks
  EORTC-QLQ-LC29 measuring the quality of life in patients with lung cancer. Each dimension in the scale has four response levels from not at all (1) to very much (4).
Clinical endpoint - overall survival | 16 weeks
  A series of secondary efficacy outcome measures will be evaluated based on overall survival from the date of the first study treatment and changes in objective response using RECIST (1.1) or iRECIST criteria. The assessed parameters will be:
  Overall Survival (OS). Overall survival ( OS ) is defined as the time from randomization to death from any cause, is a direct measure of clinical benefit to a patient.
Clinical endpoint - progression free survival | 16 weeks
  A series of secondary efficacy outcome measures will be evaluated based on overall survival from the date of the first study treatment and changes in objective response using RECIST (1.1) or iRECIST criteria. The assessed parameters will be:
  Progression Free Survival (PFS) Progression-free survival ( pfs ) is defined as time from randomization until first evidence of tumour progression or until death from any cause, whichever comes first.
Clinical endpoint - disease control rate | 16 weeks
  A series of secondary efficacy outcome measures will be evaluated based on overall survival from the date of the first study treatment and changes in objective response using RECIST (1.1) or iRECIST criteria. The assessed parameters will be:
  Disease Control Rate (DCR) Overall response rate (ORR) is defined as the proportion of patients who have a partial or complete response to therapy; it does not include stable disease and is a direct measure of drug tumoricidal activity. In contrast, disease control rate is a composite of ORR and stable disease and is useful to measure the efficacy of therapies that have tumoristatic effects rather than tumoricidal effects.
Nutritional status assessment | 16 weeks
  The Scored Patient-Generated Subjective Global Assessment (PG-SGA©) scale will be used. The Scored PG-SGA© includes the four patient-generated historical components (Weight History, Food Intake, Symptoms and Activities and Function - also known as the PG-SGA Short Form©), the professional part (Diagnosis, Age, Metabolic stress, and Physical Exam), the Global Assessment (A = well nourished, B = moderately malnourished or suspected malnutrition, C = severely malnourished) and the total numerical score.
Physical performance status assessment with 6 minute walk test (6MWT) | 16 weeks
  The physical performance assessment will be measured with 6-minute walk test (6MWT).
  6MWT meassures the distance patient covers when walking in a regular pace in standardized condition. The longer distance is expected in patients who improve while the poor patient performance and capability, the shorter distance will be measured.
Muscle performance assessment with a hand grip test | 16 weeks
  The muscle performance assessment will be measured hand grip test. The purpose of this test is to measure the maximum isometric strength of the hand and forearm muscles. The participant will be asked to squeeze the dynamometer as hard as possible with each of his or her hands in a standing position. The subject squeezes the dynamometer with maximum isometric effort, which is maintained for about 5 seconds. Results for left and right hand separately are recorded in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Ostrowski, MD, Study Director — Immunicom Inc
Locations (3):
- Turkey (Türkiye) (3):
  - Acibadem Atakent Hospital, Medical Oncology Department, Istanbul, Kucukcekmece
  - Acibadem Maslak Hospital, Medical Oncology Department - coordinating site, Istanbul, Sariyer
  - Acibadem Altunizade Hospital, Mecical Oncology Department, Istanbul, Uskudar

IPD SHARING:
Plan to Share IPD: No